CLINICAL TRIAL: NCT01198444
Title: Prospective, Open-label Observational Survey Evaluating Patients Compliance to Administration Regimen During Low Dose Combined Oral Contraceptive Use in Everyday Praxis Data on Oral Contraceptives Compliance - DOC Study
Brief Title: To Evaluate Compliance to Treatment Regimen (Rate of Deviations From the Prescribed Regimen) in Polish Females Treated With Different Low Dose Oral Contraceptives
Acronym: DOC
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Sp. z o.o.
Other Study IDs: 14340; YA0712PL (Other: Company Internal)
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Contraception
Keywords: Contraception; Compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: EE/DRSP (Yasmin Product Family)

INTERVENTIONS:
Drug: EE/DRSP (Yasmin Product Family) — One tablet per day, orally, 21 tablets followed by 7 days, during three consecutive cycles.

SUMMARY:
Adherence to the dosing scheme is the principal element of Combined Oral Contraceptives efficiency. On the other hand noncompliance seemed to be an inseparable element of any oral treatment. The aim of the study is to evaluate in everyday practice the relation between dosage errors and indicated factors, potentially influencing the compliance with the dosing scheme.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the age of over 18 requiring contraception. The decisions would be made at the discretion of the attending physician.

Exclusion Criteria:

* According to official Summary of Product Characteristics (SmPC) contraindications.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Gynecological practices patients - starters or current users.
Sampling Method: Probability Sample
Enrollment: 11884 (Actual)
Dates: Start 2007-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The percentage of users showing noncompliant behaviors | 3 consecutive cycles

SECONDARY OUTCOMES:
The characteristics of noncompliant behavior | 3 consecutive cycles
The relation between noncompliant behavior and selected factors | 3 consecutive cycles

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Poland